CLINICAL TRIAL: NCT01901523
Title: Phase II Study of Response of Medical Journal Editorial Boards to Notification of Serious Discrepancies in Published Clinical Trials in Human Patients.
Brief Title: Coordinated Assessment of Notifications of Trials Containing Overt Published Errors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Principal Investigator, Darrel Francis, Professor of Cardiology, Imperial College London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ICCH/13/SFI/Str
Record Dates: First submitted 2013-07-12; First posted 2013-07-17 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Heart Failure
Keywords: Discrepancy; Committee on Publication Ethics; Correction; Erratum; Retraction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Provision of information (Experimental): Reporting of discrepancy to journal
  Interventions: Behavioral: Reporting of discrepancy to journal

INTERVENTIONS:
Behavioral: Reporting of discrepancy to journal
  Other Names: Mathematical impossibility; Factual impossibility; Contradiction; Arithmetical impossibility; Error; Discrepancies; Fractional patients; Impossible percentage; Contradictory data; Negative standard deviation; Negative NYHA

SUMMARY:
Clinical research, like all science, is self-correcting, with errors detected by the scientific community and communicated to the publishing journals, which then relay the information (and its resolution) to its readers. If this relaying process fails, science grinds to a halt. In this study we are testing its integrity.

DETAILED DESCRIPTION:
This prospective study documents the outcome of notification to journal editorial boards (or equivalent authorities) of factually incorrect or inconsistent claims, in reports they have published.

ELIGIBILITY:
Inclusion Criteria:

* Report of a clinical trial in humans of treatment of heart disease with bone marrow derived stem cells
* Report containing discrepancy by reference to same report or another report

Exclusion Criteria:

* Discrepancy has already been corrected by an erratum

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Time to correction, retraction, or other notification to the readership of discrepancy | 12 months

SECONDARY OUTCOMES:
Time to initial response from journal | 0-4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Darrel P Francis, MA MD FRCP, Study Chair — Imperial College London
Locations (1):
- International Centre for Circulatory Health, London, London, United Kingdom

REFERENCES:
- [Background] Francis DP, Mielewczik M, Zargaran D, Cole GD. Autologous bone marrow-derived stem cell therapy in heart disease: discrepancies and contradictions. Int J Cardiol. 2013 Oct 9;168(4):3381-403. doi: 10.1016/j.ijcard.2013.04.152. Epub 2013 Jul 2. PMID 23830344
- [Background] Nowbar AN, Mielewczik M, Karavassilis M, Dehbi HM, Shun-Shin MJ, Jones S, Howard JP, Cole GD, Francis DP; DAMASCENE writing group. Discrepancies in autologous bone marrow stem cell trials and enhancement of ejection fraction (DAMASCENE): weighted regression and meta-analysis. BMJ. 2014 Apr 28;348:g2688. doi: 10.1136/bmj.g2688. PMID 24778175
- See also: Reliable cardiovascular research — http://www1.imperial.ac.uk/medicine/people/d.francis/